CLINICAL TRIAL: NCT00664248
Title: A Clinical Study Evaluating the Safety and Efficacy of IDP-110 in Patients With Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dow Pharmaceutical Sciences (Industry)
Responsible Party: Barry M. Calvarese, MS / Vice President, Regulatory & Clinical Affairs, Dow Pharmaceutical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DPSI-06-22-2006-012
Record Dates: First submitted 2008-04-15; First posted 2008-04-22 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin; Benzoyl Peroxide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: IDP-110
- 2 (Active Comparator)
  Interventions: Drug: Clindamycin
- 3 (Active Comparator)
  Interventions: Drug: Benzoyl peroxide
- 4 (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: IDP-110 — Topical application for 12 weeks
  Arms: 1
Drug: Clindamycin — Topical application for 12 weeks
  Arms: 2
Drug: Benzoyl peroxide — Topical application for 12 weeks
  Arms: 3
Drug: Vehicle — Topical application for 12 weeks
  Arms: 4

SUMMARY:
The purpose of this study is to assess the effectiveness of IDP-110 in treating patients with acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Presence of inflammatory and non-inflammatory lesions

Exclusion Criteria:

* Dermatological conditions of the face other than acne that could interfere with clinical evaluations
* Female subjects who are pregnant, nursing, planning a pregnancy, or become pregnant during the study

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1414 (Actual)
Dates: Start 2006-10; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in number of lesions | 12 weeks

SECONDARY OUTCOMES:
Change from baseline in global severity | 12 weeks

CONTACTS AND LOCATIONS:
Locations (35):
- United States (33):
  - Total Skin and Beauty Dermatology Center, Birmingham, Alabama
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - Dermatology Research of Arkansas, Little Rock, Arkansas
  - Affiliated Research Institute - Dermatology, San Diego, California
  - Therapeutics Clinical Research, San Diego, California
  - University of California, San Diego, Pediatric and Adolescent Dermatology, San Diego, California
  - Solano Clinical Research, Vallejo, California
  - Dermatology Specialists, Inc., Vista, California
  - Clinical Research Specialists, West Santa Monica, California
  - Cherry Creek Dermatology Research Inc., Denver, Colorado
  - Longmont Medical Research Network, Longmont, Colorado
  - International Dermatology Research, Inc., Miami, Florida
  - FXM Research, Miami, Florida
  - Office of Scott Glazer, MD, Buffalo Grove, Illinois
  - Henry Ford Medical Center, Detroit, Michigan
  - The Nevada Center for Dermatology, Reno, Nevada
  - Academic Dermatology, Albuquerque, New Mexico
  - Triangle Medical Research Associates, Cary, North Carolina
  - Unifour Medical Research Associates, Hickory, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - New Haven Medical Research, Wilmington, North Carolina
  - Northwest Cutaneous Research Specialists, Portland, Oregon
  - Oregon Medical Center, PC, Portland, Oregon
  - Rivergate Dermatology, Goodlettsville, Tennessee
  - Dermatology Associates, Knoxville, Tennessee
  - Dermatology Research Associates, Nashville, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - The Center for Skin Research, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Dermatology Resarch Center, Salt Lake City, Utah
  - Advanced Clinical Research - Jordan Valley, West Jordan, Utah
  - Advanced Healthcare, Milwaukee, Wisconsin
- Dermatology and Skin Surgery Centre, Belize City, Belize
- Mediprobe Research, New London, Ontario, Canada